CLINICAL TRIAL: NCT02228668
Title: Follow up to the AVANT Study up to 8 and 10 Years (Median Follow up) in Patients With Colon Carcinoma
Status: Completed | Type: Observational
Sponsor: GERCOR - Multidisciplinary Oncology Cooperative Group (Other)
Collaborators: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: S-AVANT C13-1
Record Dates: First submitted 2014-08-08; First posted 2014-08-29 (Estimated); Last update posted 2019-02-27 (Actual); Status verified 2019-02

CONDITIONS: Colon Cancer Treated With Bevacizumab After Colon Surgery
Keywords: AVANT; GERCOR; Follow up; Colon cancer; Bevacizumab; Overall survival
MeSH Terms: conditions — Colonic Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Other
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of the S-AVANT study is to collect additional data at 8 and 10 years median follow up of patients previously included in the AVANT trial from December 2004 to June 2007.

Clinical data of the AVANT trial will be updated. Neither additional examination nor administration of any treatment will be performed on the patients.

330 centers in 34 countries participated to the AVANT trial (Australia, Austria , Belgium, Brazil, Bulgaria, Canada, China/Hong-Kong, Czeck Republic, Finland, France, Germany, Greece, Hungary, Israël, Italy, Japan, Korean Republic, Mexico, Netherlands, New Zealand, Norway, Panama, Poland, Portugal, Russia Federation, Singapore, South Africa, Spain, Sweden, Switzerland, Taïwan, Thaïland, United Kingdom, U.S.A).

The AVANT study aiming at demonstrating superiority of bevacizumab in combination with FOLFOX-4 or XELOX compared to FOLFOX-4, did not show prolongation of DFS at 3 year when adding bevacizumab to chemotherapy in resected stage III colon cancer.

Adverse events were consistent with the known safety profile of bevacizumab. However, more relapses and deaths due to disease progression have been observed in both bevacizumab arms.

A more prolonged follow-up is necessary to assess overall survival and to evaluate long-term results and safety.

Collection of additional follow-up data will start Q3 2014. Clinical data are to be collected at 8-year median follow-up (expected to be reached around Q2 2014) and at 10-year median follow-up (expected to be reached around Q2 2016).

All analyses will be performed on an exploratory purpose only. An analysis at 8 years median follow-up and a final analysis at 10 years median follow-up will be performed in the main population (all randomized patients in the AVANT trial including patients lost to follow up or died).

ELIGIBILITY:
Inclusion Criteria:

* All patients randomized in the AVANT trial.

Exclusion Criteria:

* Written opposition from alive patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with colon cancer included in the AVANT trial and who were randomized between the three arms of treatment:
  * ARM A: (FOLFOX-4): Oxaliplatin, leucovorin (LV) and 5-fluorouracil (5-FU).
  * ARM B: (FOLFOX-4+bev): Bevacizumab, oxaliplatin, leucovorin (LV) and 5-fluorouracil (5-FU).
  * ARM C: (XELOX+ bev): Bevacizumab, oxaliplatin in combination with capecitabine.
Sampling Method: Non-Probability Sample
Enrollment: 1636 (Actual)
Dates: Start 2015-03; Primary Completion 2019-02-15 (Actual); Study Completion 2019-02-15 (Actual)

PRIMARY OUTCOMES:
Overall Survival (OS) up to 8 and 10 years median follow-up of the stage III population randomized in the AVANT study. | From randomization until 10 years median follow-up, assessed up to 5 years from the beginning of the S-AVANT study.

SECONDARY OUTCOMES:
Overall Survival (OS) in stage III patients at 8 years median follow-up in the subgroup of alive patients not lost to follow-up after the AVANT trial ending. | From randomization until 8 years median follow-up, assessed up to 3 years from the beginning of the S-AVANT study.
Disease-Free Survival (DFS) in stage III patients at 8 and 10 years median follow-up. | From randomization until 10 years median follow-up, assessed up to 5 years from the beginning of the S-AVANT study.
Relapse Free Survival (RFS) in patients with stage II and stage III colon cancer. | From randomization until first relapse, assessed up to 5 years from the beginning of the S-AVANT study.
Cancer Specific Survival (CSS) in patients with stage II and stage III colon cancer. | From randomization until the date of death related to primary cancer or second primary colon cancer, assessed up to 5 years from the beginning of the S-AVANT study.

CONTACTS AND LOCATIONS:
Overall Officials: Aimery de Gramont, Pr, Study Director — GERCOR - Multidisciplinary Oncology Cooperative Group
Locations (1):
- GERCOR, Paris, France

REFERENCES:
- [Derived] Chibaudel B, Henriques J, Rakez M, Brenner B, Kim TW, Martinez-Villacampa M, Gallego-Plazas J, Cervantes A, Shim K, Jonker D, Guerin-Meyer V, Mineur L, Banzi C, Dewdney A, Dejthevaporn T, Bloemendal HJ, Roth A, Moehler M, Aranda E, Van Cutsem E, Tabernero J, Schmoll HJ, Hoff PM, Andre T, de Gramont A. Association of Bevacizumab Plus Oxaliplatin-Based Chemotherapy With Disease-Free Survival and Overall Survival in Patients With Stage II Colon Cancer: A Secondary Analysis of the AVANT Trial. JAMA Netw Open. 2020 Oct 1;3(10):e2020425. doi: 10.1001/jamanetworkopen.2020.20425. PMID 33074326
- See also: Related Info — http://www.thelancet.com/journals/lanonc/article/PIIS1470-2045(12)70509-0/abstract